CLINICAL TRIAL: NCT04228926
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of ZKY001 Eye Drops in Patients With Corneal Epithelial Defects After Corneal Endothelial Transplantation
Brief Title: Evaluating the Efficacy and Safety of ZKY001 Eye Drops in the Treatment of Corneal Epithelial Defects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZK-SFT-2019
Record Dates: First submitted 2020-01-01; First posted 2020-01-14 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Corneal Defect

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.002% ZKY001 eye drops (Experimental): Experimental group A: 35 subjects .0.002% ZKY001 eye drops . 4 times a day,1 drop every time, continuously administered for 14±2 days ZKY001 eye drops will be directly dripped into the test eye (the surgical eye was taken as the test eye).
  Interventions: Drug: ZKY001 eye drops 0.3g:0.006mg
- 0.004% ZKY001 eye drops (Experimental): Experimental group B: 35 subjects .0.004% ZKY001 eye drops . 4 times a day,1 drop every time, continuously administered for 14±2 days ZKY001 eye drops will be directly dripped into the test eye (the surgical eye was taken as the test eye).
  Interventions: Drug: ZKY001 eye drops 0.3g:0.012mg
- The placebo (Placebo Comparator): Placebo group C: ZKY001 simulated eye drops .4 times a day,1 drop every time, continuously administered for 14±2 days ZKY001 simulated eye drops will be directly dripped into the test eye (the surgical eye was taken as the test eye).
  Interventions: Drug: ZKY001 simulated eye drops

INTERVENTIONS:
Drug: ZKY001 eye drops 0.3g:0.006mg — ZKY001 eye drops of 0.002% continuously for up to 14±2 days after Corneal endothelial transplantation
  Other Names: shengfatai-eye drops; the Germinal Peptide eye drops
  Arms: 0.002% ZKY001 eye drops
Drug: ZKY001 eye drops 0.3g:0.012mg — ZKY001 eye drops of 0.004% continuously for up to 14±2 days after Corneal endothelial transplantation
  Other Names: shengfatai-eye drops; the Germinal Peptide eye drops
  Arms: 0.004% ZKY001 eye drops
Drug: ZKY001 simulated eye drops — ZKY001 simulated eye drops continuously for up to 14±2 days after Corneal endothelial transplantation
  Other Names: the placebo
  Arms: The placebo

SUMMARY:
The subjects of this study were patients who underwent corneal endothelial transplantation,who were randomly divided into 3 groups, 2 groups (0.002% and 0.004% ZKY001 eye drops) and 1 placebo control group.

DETAILED DESCRIPTION:
This study is an exploratory phase II clinical study with no sample size estimation.According to the results of the preliminary animal experiments and phase I clinical trials, 2 concentrations (0.002% and 0.004%ZKY001eye drops) were selected as the experimental group, and 1 placebo control group was selected, with 35 subjects in each group and a total of 105 subjects.Each subject will drop the study drug into the test eye (the surgical eye is taken as the test eye) according to the randomly assigned drug number.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-80, regardless of gender;
2. patients who have undergone DSAEK or DMEK and need to remove corneal epithelium;
3. Schirmer test I ≥10mm/5min;
4. normal corneal limbus structure under slit lamp during screening period;
5. sign the informed consent.

Exclusion Criteria:

1. intraocular pressure > 21mmHg or baseline intraocular pressure > 35mmHg during screening period;
2. fasting blood glucose > 9.0mmol/L during screening period;
3. postoperative complications occurred, such as dislocation of the implant and high intraocular pressure caused by air bubbles in the anterior chamber;
4. suffered from eye infection, optic neuritis, pigment membrane inflammation, or fundus, macular lesions that affect vision, glaucoma;
5. serious cardiovascular history (congestive heart failure, uncontrolled hypertension, unstable coronary heart disease or myocardial infarction or severe arrhythmia, etc.);
6. severe hepatic and renal insufficiency, alanine aminotransferase (ALT), alanine aminotransferase (AST) ≥ 2 times the normal upper limit, blood creatinine (Cr) ≥ 1.5 times the normal upper limit;
7. those who wear contact lenses within 3 days before screening;
8. screening drugs that have used corneal repair effect within the first 3 days;
9. have received corneal refractive surgery or keratoplasty;
10. have received internal eye surgery within 3 months before screening or need to undergo internal eye surgery during the study period;
11. have participated in other clinical trials or are participating in other clinical trials within 3 months prior to screening;
12. suffering from central nervous system disease and/or mental state inability to cooperate;
13. women in pregnancy, lactation or childbearing age do not take effective contraceptive measures;
14. allergy to the test product and basic drugs;
15. patients who are not considered appropriate to participate in this study, including those who are unable or unwilling to comply with the protocol requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-12-24 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of corneal epithelial defect area on Day 3 compared with that on baseline will be calculated by the grid method | Day 3, 8:00 am±1hour
  Subjects will undergo fluorescein staining of the cornea, slit-lamp examination and photography (8:00 ±1h) before first administration on Day1（the first day after surgery,baseline），Day3 (the third day after surgery).After slit-lamp photography was scanned by the scanner, image pro plus software was used to scale the photo to the same size as the test eye, and then the grid method was used to calculate the area of the corneal defect in the photo.
  Improvement in epithelial defect area = defect area on baseline - defect area on Day3

SECONDARY OUTCOMES:
The subject's symptoms and signs will be evaluated on the General Arbitroid | Day 3, Day6 、Day15 8:00 am±1hour
  Subjects' symptoms and signs were evaluated on the general symptom and signs scale at Day1 before fluorescein staining of the cornea.
  The mean change of the total score of symptoms and signs on Day 3、Day6 、Day15 after the operation compared with the baseline
Scoring with D6 and D15 corneal fluorescein staining | Day6 、Day15 8:00 am±1hour
  Subjects underwent corneal fluorescein staining and scoring before the first dose of Day1, Day6 and Day15
The improvement rate of corneal epithelial defect area on Day 3 postoperation after surgery compared with that at baseline (Day1 postoperation ) will be calculated by the grid method | Day 3, 8:00 am±1hour
  Subjects will undergo fluorescein staining of the cornea, slit-lamp examination and photography (8:00 ±1h) before first administration on Day1（the first day after surgery,baseline），Day3 (the third day after surgery).After slit-lamp photography was scanned by the scanner, image pro plus software was used to scale the photo to the same size as the test eye, and then the grid method was used to calculate the area of the corneal defect in the photo.
  Improvement rate of corneal epithelial defect area=( defect area at baseline - defect area at Day3)/defect area at baseline ✖100%
The change of corneal epithelial defect area on Day 2、Day4、Day5 compared with that on baseline(Day 1) will be calculated by the grid method | Day 2、Day4、Day5 8:00 am±1hour
  Subjects will undergo fluorescein staining of the cornea, slit-lamp examination and photography (8:00 ±1h) before first administration on Day1，Day 2、Day4、Day5.After slit-lamp photography was scanned by the scanner, image pro plus software was used to scale the photo to the same size as the test eye, and then the grid method was used to calculate the area of the corneal defect in the photo.
  Day2 Improvement in epithelial defect area = defect area on baseline - defect area on Day2
  Day4Improvement in epithelial defect area = defect area on baseline - defect area on Day4
  Day5 Improvement in epithelial defect area = defect area on baseline - defect area on Day5
The incidence of reexfoliation of corneal epithelium was observed | Day 3, Day4，Day5，Day6，Day15±2 8:00 am±1hour
  incidence of re-exfoliation of corneal epithelium on Day3、Day4、Day5、Day6、Day15±2 In the process of corneal epithelium repair, the epithelium may reexfoliate after covering the wound.Reexfoliation of the corneal epithelium was defined as positive corneal fluorescein staining under slit lamp microscope，Corneal fluorescein staining was performed before the first administration

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zhao, PHD, Study Director — Beijing Tongren Hospital
Locations (1):
- Eye ＆ Ent Hospital of Fudan University, Shanghai, Shanghai Municipality, China